CLINICAL TRIAL: NCT02149329
Title: Short Versus Extended Antibiotic Treatment With a Carbapenem for High-risk Febrile Neutropenia in Hematology Patients With Fever of Unknown Origin: a Randomized Multicenter Non-inferiority Trial.
Brief Title: Short Versus Extended Antibiotic Treatment With a Carbapenem for High-risk Febrile Neutropenia in Hematology Patients With FUO
Acronym: SHORT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); FondsNutsOhra (Unknown)
Responsible Party: Principal Investigator, Nick de Jonge, MD, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000735; 2014-001546-25 (EudraCT Number); NL48960.029.14 (Registry Identifier: CCMO (Nationale research committee) file number)
Record Dates: First submitted 2014-05-19; First posted 2014-05-29 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Febrile Neutropenia; Hematological Malignancy
Keywords: fever; neutropenia; febrile neutropenia; carbapenem; imipenem; meropenem; antibiotic stewardship; hematology; oncology
MeSH Terms: conditions — Febrile Neutropenia; Hematologic Neoplasms; Fever; Neutropenia; Neoplasms | interventions — Meropenem; Cilastatin, Imipenem Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Short treatment (Experimental): Discontinuation of imipenem-cilastatin or meropenem after 3x24 hours irrespective of presence of fever.
  Interventions: Drug: Discontinuation of imipenem-cilastatin or meropenem
- Extended treatment (No Intervention): Extended treatment with imipenem-cilastatin or meropenem for at least 6 more days. The treatment with a carbapenem will be continued until patients have been treated for at least 9x24 hours and have been afebrile (tympanic membrane temperature <38.0°C) for at least five consecutive days or until resolution of neutropenia (ANC > 0,5 x10^9/L), whichever comes first.

INTERVENTIONS:
Drug: Discontinuation of imipenem-cilastatin or meropenem — Discontinuation of imipenem-cilastatin or meropenem after 3x24 hours irrespective of presence of fever.
  Other Names: tienam (imipenem-cilastatin)
  Arms: Short treatment

SUMMARY:
A multicenter open-label non-inferiority randomized clinical trial comparing the safety (non-inferiority) of short antibiotic treatment (72 hours) with an anti-pseudomonal carbapenem with regard to treatment failure in comparison with extended treatment (at least 9 days) of high-risk febrile neutropenia in hematology patients receiving standard antimicrobial prophylaxis.

DETAILED DESCRIPTION:
Episodes of fever are very common in patients undergoing intensive chemotherapy treatment for malignant hematological disease. More than 80% of patients experience one or more episodes of fever after their first cycle of chemotherapy. Only 20-30% of these patients have a clinically documented focus and mostly include infections of skin, intestinal tract and lung, while at most 10-25% of these patients have microbiologically proven bacteremia during these episodes. Patients with malignant hematological diseases and intensive chemotherapy induced neutropenia are extremely prone to overwhelming bacterial infections. Therefore, empirical antibiotic treatment is initiated at the first occurrence of fever, even if no apparent cause for the fever is evident. Most protocols advice treatment with very broad-spectrum antibiotics, mostly anti-pseudomonal carbapenems or fourth generation anti-pseudomonal cephalosporins.

Prolonged continuation of treatment may induce bacterial resistance. In view of the possible emergence of bacterial resistance due to prolonged antibiotic administration, continuation until recovery of neutropenia is suboptimal because it is costly because of longer hospital admissions, higher antibiotics costs and more possible adverse reactions.

Recent observational data (Slobbe et al) has showed that in adult hematological patients with febrile neutropenia, discontinuation of empiric antibacterial therapy after three days can be safe if no infectious etiology can be found, even in cases with persistent fever. However no RCT has hitherto been performed to support this observational data.

This study compares the safety (non-inferiority) of short treatment (72 hours) versus extended treatment (at least 9 days) with an anti-pseudomonal carbapenem for hematology patients with unexplained high risk febrile neutropenia. We hypothesize that a more restrictive use of broad-spectrum antibiotic use of three days in unexplained fever in neutropenic hematology patients is non-inferior to the present extended use during at least 9 days which would lead to a more restrictive use of antibiotics and less multiresistant strains of bacteria, costs and hospitalization length in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with malignant hematological diseases being treated with cytotoxic chemotherapy or stem cell transplantation;
2. High-risk neutropenia (Absolute neutrophil count (ANC) <0.5x109/L which is expected to last longer than 7 days);
3. Fever (One single measured tympanic membrane temperature of >38.5°C or a temperature of >38.0°C during 2 subsequent measurements separated by at least 2 hours);
4. Age 18 years or older;
5. Written informed consent.

Exclusion Criteria:

1. Contraindications to use of imipenem-cilastatin or meropenem such as allergy, previous severe side-effects or previous microbiological cultures with carbapenem-resistant microorganism(s).
2. Corticosteroid use ≥10 mg per day prednisolone or equivalent for more than 3 consecutive day during the previous 7 days.
3. Clinically or microbiologically documented infection.
4. Symptoms of septic shock (systolic blood pressure <90 mm Hg unresponsive to fluid resuscitation and/or oliguria (urine production <500mL/day).
5. Previous enrollment in this study during the same episode of neutropenia.
6. Any critical illness for which Intensive Care Unit treatment is required.
7. Legal incompetency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2019-08-05 (Actual); Study Completion 2019-08-05 (Actual)

PRIMARY OUTCOMES:
The percentage of patients with failed treatment | Between randomization (at 3x24 hours) and before 9x24hours after treatment initiation)
  Treatment failure is defined as the occurrence of one of the following events after 3x24 hours and before 9x24hours after treatment initiation with a carbapenem:
  -A clinically or microbiologically documented carbapenem-sensitive infection; treatment.
  Recurrence of fever after previous defervescence (tympanic temperature <38.0 °C during 24 hours) which is not attributable to administration of a blood product or to a drug reaction.
  o In case of clinical doubt whether the fever is of infectious etiology, the recurrence of fever will be considered as failure.
Death/ARDS or Septic shock | From randomization until the end of neutropenia (neutrophil count >=0.5x10e9/L) up to 6 months after randomization.
  The occurrence of death, ARDS/respiratory insufficiency, septic shock (systolic blood pressure <90 mmHg and oliguria <500 mL/day) due to any cause.

SECONDARY OUTCOMES:
All-cause mortality. | 1. From 3x24hours of treatment until the end of neutropenia. 2. Within 30 days after the end of neutropenia
Infection-related mortality. | 1. From 3x24hours of treatment until the end of neutropenia. 2.Within 30 days after recovery of neutropenia
The length of hospitalization in days. | From admission until discharge, with an estimated average of 4 weeks
Treatment strategy failure | after 3x24hours of treatment with a carbapenem and until the end of the neutropenic episode
  Treatment strategy failure is defined as occurrence of any of the following events after 3x24hours of treatment with a carbapenem and until the end of the neutropenic episode:
  1. Any clinically or microbiologically documented infection.
  2. The recurrence of fever after previous defervescence during neutropenia.
  3. Death, septic shock or ARDS/respiratory failure due to any cause
  4. Adverse drug-related events due to a carbapenem requiring (temporary) interruption of treatment, including but not exclusively: liver and kidney dysfunction, convulsion and allergic reactions.
  5. Unexpected re-admission within 30 days after discharge other than for planned chemotherapy or other elective treatment.
  6. Antibiotic or antifungal treatment within 30days after discharge other than standard antibiotic prophylaxis.
The total number of febrile episodes during neutropenia. | From the start of neutropenia (ANC<0.5x10^9) until the end of neutropenia, an expected average of 21 days
Time to defervescence | Onset of fever until defervenscence, an expected average of 5 days.
  Fever is defined as one single measured tympanic membrane temperature of >38.5°C or a temperature of >38.0°C during 2 subsequent measurements separated by at least 2 hours.
  Defervescence is defined as three times a tympanic membrane temperature <37.5 °C with a minimal measurement interval of at least 8 hours
Incidence and prevalence of Clostridium difficile infection | Onset of fever until 30 days after the end of neutropenia.
Candida spp. colonization in (surveillance) cultures | From onset of fever until 30 days after the end of neutropenia.
Cost of antimicrobial therapy per admission | From admission until discharge, with an estimated average of 4 weeks
The percentage of patients with a MASCC-score≥21 and treatment failure (defined as in primary endpoint) | From the onset of fever until the end of the neutropenic episode, with an estimated average of 21 days.
The percentage of patients with mucositis and positive blood cultures or short treatment failure. | From onset of fever until 30 days after end of neutropenia.
Bacterial resistance in blood cultures and surveillance cultures (including minimal inhibitory concentrations (MIC)). | All previous cultures and cultures performed until 30 days after the end of neutropenia.
The incidence and prevalence of fungal, viral, or carbapenem-resistant (inherent/acquired) infections until the end of neutropenia | om the onset of fever until the end of the neutropenic episode, with an estimated average of 21 days.
Late treatment failure | Between 9x24hours and 14x24hours after onset of treatment with a carbapemen.
  Defined as primary endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen JWM Janssen, MD, PhD, Principal Investigator — Amsterdam UMC, location VUmc; Michiel A van Agtmael, MD, PhD, Principal Investigator — Amsterdam UMC, location VUmc; Mark MH Kramer, Prof., MD, Study Chair — Amsterdam UMC, location VUmc; Sonja Zweegman, Prof.,MD, Study Chair — Amsterdam UMC, location VUmc
Locations (2):
- Netherlands (2):
  - VU university medical center, Amsterdam
  - HAGA ziekenhuis, The Hague

REFERENCES:
- [Derived] de Jonge NA, Janssen JJWM, Ypma P, Herbers AHE, de Kreuk A, Vasmel W, van den Ouweland JMW, Beeker A, Visser O, Zweegman S, Blijlevens NMA, van Agtmael MA, Sikkens JJ. Mucositis-associated bloodstream infections in adult haematology patients with fever during neutropenia: risk factors and the impact of mucositis severity. Support Care Cancer. 2024 Aug 8;32(9):579. doi: 10.1007/s00520-024-08776-w. PMID 39115709
- [Derived] de Jonge NA, Sikkens JJ, Zweegman S, Beeker A, Ypma P, Herbers AH, Vasmel W, de Kreuk A, Coenen JLLM, Lissenberg-Witte B, Kramer MHH, van Agtmael MA, Janssen JJWM. Short versus extended treatment with a carbapenem in patients with high-risk fever of unknown origin during neutropenia: a non-inferiority, open-label, multicentre, randomised trial. Lancet Haematol. 2022 Aug;9(8):e563-e572. doi: 10.1016/S2352-3026(22)00145-4. Epub 2022 Jun 9. PMID 35691326